CLINICAL TRIAL: NCT03732677
Title: A Phase III, Randomized, Open-Label, Multi-Center, Global Study to Determine the Efficacy and Safety of Durvalumab in Combination With Gemcitabine+Cisplatin for Neoadjuvant Treatment Followed by Durvalumab Alone for Adjuvant Treatment in Patients With Muscle-Invasive Bladder Cancer.
Brief Title: Durvalumab+ Gemcitabine/Cisplatin (Neoadjuvant Treatment) and Durvalumab (Adjuvant Treatment) in Patients With MIBC
Acronym: NIAGARA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D933RC00001; 2023-510015-19-00 (Registry Identifier: CTIS); 2018-001811-59 (EudraCT Number)
Record Dates: First submitted 2018-10-05; First posted 2018-11-06 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Muscle Invasive Bladder Cancer
Keywords: Bladder Cancer; Immunotherapy; PD-L1; Durvalumab (MEDI4736)
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Chemotherapy + Durvalumab
  Interventions: Drug: Durvalumab; Drug: Cisplatin; Drug: Gemcitabine
- Arm 2 (Active Comparator): Chemotherapy alone
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Durvalumab — Anti- PD-L1 Antibody
  Arms: Arm 1
Drug: Cisplatin — Chemotherapy Agent
Drug: Gemcitabine — Chemotherapy agent

SUMMARY:
A Global Study to Determine the Efficacy and Safety of Durvalumab in Combination with Gemcitabine+Cisplatin for Neoadjuvant Treatment and Durvalumab Alone for Adjuvant Treatment in Patients with Muscle-Invasive Bladder Cancer

ELIGIBILITY:
Inclusion:

* Patient resectable muscle-invasive bladder cancer with clinical stage T2-T4aN0/1M0 with transitional and mixed transitional cell histology
* Patients must be planning to undergo a radical cystectomy
* Patients who have not received prior systemic chemotherapy or immunotherapy for treatment of MIBC
* ECOG performance status of 0 or 1
* Must have a life expectancy of at least 12 weeks at randomization

Exclusion:

* Evidence of lymph node (N2-N3) or metastatic (M1) disease at time of screening.
* Prior pelvic radiotherapy treatment within 2 years of randomization to study
* Prior exposure to immune-mediated therapy (with exclusion of Bacillus-Calmette Guerin [BCG]), including but not limited to other anti-CTLA-4, anti-PD-1, anti PD-L1, or anti-PD-L2 antibodies.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of investigational product (IP). The following are exceptions to this criterion: Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection); Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent; Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.
* Uncontrolled intercurrent illness
* Active infection including Tuberculosis, Hepatitis B, Hepatitis C, and Human Immunodeficiency

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1063 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (162):
- United States (18):
  - Research Site, Birmingham, Alabama
  - Research Site, Los Angeles, California
  - Research Site, Palo Alto, California
  - Research Site, New Haven, Connecticut
  - Research Site, Chicago, Illinois
  - Research Site, Geneva, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Westwood, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Towson, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Burlington, Vermont
  - Research Site, Milwaukee, Wisconsin
- Australia (6):
  - Research Site, Brisbane
  - Research Site, Elizabeth Vale
  - Research Site, Macquarie University
  - Research Site, Melbourne
  - Research Site, Murdoch
  - Research Site, South Brisbane
- Belgium (6):
  - Research Site, Bruges
  - Research Site, Charleroi
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Roeselare
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santa Maria
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (7):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
- Chile (5):
  - Research Site, Antofagasta
  - Research Site, Port Montt
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- France (8):
  - Research Site, Angers
  - Research Site, Dijon
  - Research Site, Grenoble
  - Research Site, Montpellier
  - Research Site, Nîmes
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Rouen
- Germany (15):
  - Research Site, Bergisch Gladbach
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Erlangen
  - Research Site, Göttingen
  - Research Site, Herne
  - Research Site, Jena
  - Research Site, Magdeburg
  - Research Site, Mannheim
  - Research Site, Münster
  - Research Site, Nuremberg
  - Research Site, Oldenburg
  - Research Site, Regensburg
  - Research Site, Ulm
  - Research Site, Würzburg
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Italy (8):
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Pozzuoli
  - Research Site, Verona
- Japan (17):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hirosaki-shi
  - Research Site, Hiroshima
  - Research Site, Kanazawa
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Miyazaki
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sendai
  - Research Site, Toyama
  - Research Site, Tsukuba
  - Research Site, Yokohama
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Rotterdam
- Philippines (6):
  - Research Site, Baguio City
  - Research Site, Cebu
  - Research Site, Davao City
  - Research Site, Makati
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (10):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Grudziądz
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Ostrołęka
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (8):
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Ufa
  - Research Site, Vologda
- South Korea (5):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Seoul
- Spain (7):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Santander
  - Research Site, Seville
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Karşıyaka
- United Kingdom (5):
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Nottingham
  - Research Site, Sheffield
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Powles T, Catto JWF, Galsky MD, Al-Ahmadie H, Meeks JJ, Nishiyama H, Vu TQ, Antonuzzo L, Wiechno P, Atduev V, Kann AG, Kim TH, Suarez C, Chang CH, Roghmann F, Ozguroglu M, Eigl BJ, Oliveira N, Buchler T, Gadot M, Zakharia Y, Armstrong J, Gupta A, Hois S, van der Heijden MS; NIAGARA Investigators. Perioperative Durvalumab with Neoadjuvant Chemotherapy in Operable Bladder Cancer. N Engl J Med. 2024 Nov 14;391(19):1773-1786. doi: 10.1056/NEJMoa2408154. Epub 2024 Sep 15. PMID 39282910
- See also: D933RC00001_CSR synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933RC00001&attachmentIdentifier=1bd33049-7e73-46d5-b0dc-5d91d6c5f0ef&fileName=D933RC00001_CSR_synopsis_Redacted.pdf&versionIdentifier=
- See also: D933RC00001_CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933RC00001&attachmentIdentifier=64fb18ca-1077-46c8-987e-4a5df41ef046&fileName=D933RC00001_CSP_Redacted.pdf&versionIdentifier=
- See also: D933RC00001_SAP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933RC00001&attachmentIdentifier=09d5156a-320d-4a52-92f2-c61afe4b7d9f&fileName=D933RC00001_SAP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients randomized to treatments Arm 1 or Arm 2, will be treated according to their renal function. Recruitment for borderline renal function patients will be limited to up to 20% of the targeted global population. Recruitment for patients with T2N0 disease will be limited to approximately 40% of the targeted global population; once the 40% cap has been reached, only T2-4N1M0 and T3-4N0M0 patients will be allowed to be enrolled onto the study. Completion status is reported by treatment phase
Groups:
- Durvalumab + Gemcitabine + Cisplatin: Treatments and dosing regimens: Durvalumab 1500 mg IV q3w (neoadjuvant) 1500 mg IV q4w (adjuvant post-radical cystectomy) Day 1 and Day 8 (gemcitabine 1000 mg/m2 IV) of each 21-day cycle (neoadjuvant) Day 1 and Day 8 (cisplatin 35mg/m2 IV) or Day 1 (cisplatin 70 mg/m2 IV) each 21-day cycle (neoadjuvant) Dosing will be adjusted based on renal function
- Gemcitabine + Cisplatin: Treatments and dosing regimens: Day 1 and Day 8 (gemcitabine1000 mg/m2 IV) of each 21-day cycle (neoadjuvant) Day 1 and Day 8 (cisplatin 35mg/m2 IV) or Day 1 (cisplatin 70 mg/m2 IV) each 21-day cycle (neoadjuvant) Dosing will be adjusted based on renal function
Period: Overall Study
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Started | 533 | 530
Started Neoadjuvant Treatment | 530 | 526
Completed Neoadjuvant Treatment | 417 | 389
Completed Radical Cystectomy | 469 | 441
Started Adjuvant Treatment | 383 | 0
Completed Adjuvant Treatment | 288 | 0
Completed (Completion status is reported by treatment phase) | 0 | 0
Not Completed | 533 | 530
Not completed — Terminated the study | 154 | 197
Not completed — Continuing study off treatment | 379 | 333

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin | Total
Number analyzed (Participants) | 533 | 530 | 1063
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (8.9) | 64.6 (8.9) | 64.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 97 | 193
  Male | 437 | 433 | 870
Race/Ethnicity, Customized [Number; unit: Participants]
  HISPANIC OR LATINO | 44 | 41 | 85
  MISSING | 6 | 12 | 18
  NOT HISPANIC OR LATINO | 483 | 477 | 960
Race/Ethnicity, Customized [Number; unit: Participants]
  ASIAN | 152 | 145 | 297
  BLACK OR AFRICAN AMERICAN | 6 | 4 | 10
  MISSING | 14 | 22 | 36
  OTHER | 7 | 1 | 8
  WHITE | 354 | 358 | 712

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rates at Time of Cystectomy
Description: pCR rate is defined as the proportion of patients whose pathological staging was T0N0M0 as assessed per central pathology review using specimens obtained via radical cystectomy following the neoadjuvant treatment. The denominator for pCR will be the number of patients in the FAS.
Time Frame: Up to 6 months
Population: Full Analysis Set (Intention to Treat): includes all randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 533 | 530
Participants | 199 | 146
Statistical Analysis 1: Comparison: Durvalumab + Gemcitabine + Cisplatin vs Gemcitabine + Cisplatin; Test type: Superiority; p = 0.0005, Regression, Logistic; Strata adjusted odds ratio by the logistic regression method adjusting for stratification factors: renal function , tumor stage and PDL1 status; Odds Ratio (OR) = 1.60, 95% CI 2-sided [1.227 to 2.084]

2. Primary Outcome: Event-free Survival (EFS) Per Central Review Defined as Time From Randomization to Event
Description: EFS is defined as the time from randomization to the first recurrence of disease post radical cystectomy, time of first documented progression in patients who were medically precluded for radical cystectomy, or time of expected surgery in patients who refuse to undergo a radical cystectomy or failure to undergo a radical cystectomy in participants with residual disease, or the time of death due to any cause, whichever occurs first
Time Frame: Up to 48 months
Population: The full analysis set (FAS) includes all randomized patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 533 | 530
months | NA [13.4 to NA] — Median EFS was not reached due to insufficient number of participants with events 75th percentile EFS was not reached due to insufficient number of participants with events. | 46.1 [8.6 to NA] — 75th percentile EFS was not reached due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Durvalumab + Gemcitabine + Cisplatin vs Gemcitabine + Cisplatin; Test type: Superiority; p < 0.0001, Log Rank — Stratified by renal function(adequate vs borderline),tumor stage(T2N0 vs >T2N0), PDL1 status(high vs low/negative); Hazard Ratio (HR) = 0.68, 95.877% CI 2-sided [0.554 to 0824] — The HR and CI were estimated from a stratified Cox proportional hazard model adjusting for renal function (adequate vs borderline), tumor stage (T2N0 vs >T2N0) and PDL1 status (high vs low/negative); 95% CI for hazard ratio: 0.558 - 0.817

3. Secondary Outcome: Event-free Survival at 24 Months (EFS24) Per Central Review Defined as Time From Randomization to Event
Description: EFS24 is defined as the Kaplan-Meier estimate of EFS at 24 months after randomization, as assessed per blinded independent central review or by central pathology review if a biopsy is required for a suspected new lesion, and per local investigator or local biopsy review if a biopsy is required for a suspected new lesion
Time Frame: Up to 24 months
Population: The full analysis set (FAS) Intention to treat included all randomized patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 533 | 530
Percentage of participants | 67.8 [63.6 to 71.7] | 59.8 [55.4 to 64]
Statistical Analysis 1: Comparison: Durvalumab + Gemcitabine + Cisplatin vs Gemcitabine + Cisplatin; Test type: Superiority; p = 0.0021, Chi-squared; P-value is based on a chi-squared test with one degree of freedom; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.62 to 0.90] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Proportion of Patients Who Undergo Cystectomy
Description: The proportion of patients who undergo cystectomy is defined as the proportion patients who undergo radical cystectomy after the neoadjuvant treatment. The denominator will be patients in the FAS.
Time Frame: Up to 6 months
Population: The full analysis set (FAS) Intention to treat included all randomized patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 533 | 530
Participants | 469 | 441
Statistical Analysis 1: Comparison: Durvalumab + Gemcitabine + Cisplatin vs Gemcitabine + Cisplatin; Test type: Superiority; p = 0.0265, Regression, Logistic; Stratified by renal function(adequate vs borderline),tumor stage(T2N0 vs >T2N0), PDL1 status(high vs low/negative); Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.047 to 2.095] — Strata adjusted odds ratio by the logistic regression method. Stratified by adjusting for renal function (adequate vs borderline), tumor stage (T2N0 vs >T2N0) and PDL1 status (high vs low/negative)

5. Secondary Outcome: Overall Survival
Description: OS is defined as the time from the date of randomization until death due to any cause regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy (i.e., date of death or censoring - date of randomization + 1)
Time Frame: Up to 65 months
Measure: Median (Inter-Quartile Range); unit: Months
Groups:
- Durvalumab+Gemcitabine+Cisplatin: Durvalumab + Gemcitabine + Cisplatin Treatments and dosing regimens: Durvalumab 1500 mg IV q3w (neoadjuvant) 1500 mg IV q4w (adjuvant post-radical cystectomy) Day 1 and Day 8 (gemcitabine 1000 mg/m2 IV) of each 21-day cycle (neoadjuvant) Day 1 and Day 8 (cisplatin 35mg/m2 IV) or Day 1 (cisplatin 70 mg/m2 IV) each 21-day cycle (neoadjuvant) Dosing will be adjusted based on renal function
- Gemcitabine+Cisplatin: Treatments and dosing regimens: Day 1 and Day 8 (gemcitabine1000 mg/m2 IV) of each 21-day cycle (neoadjuvant) Day 1 and Day 8 (cisplatin 35mg/m2 IV) or Day 1 (cisplatin 70 mg/m2 IV) each 21-day cycle (neoadjuvant) Dosing will be adjusted based on renal function
Arm/Group | Durvalumab+Gemcitabine+Cisplatin | Gemcitabine+Cisplatin
Number analyzed (Participants) | 533 | 530
Months | NA [41.9 to NA] — Median OS was not reached due to insufficient number of participants with events 75th percentile OS was not reached due to insufficient number of participants with events. | NA [24.1 to NA] — Median OS was not reached due to insufficient number of participants with events 75th percentile OS was not reached due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Durvalumab+Gemcitabine+Cisplatin vs Gemcitabine+Cisplatin; Test type: Superiority; p = 0.0106, Log Rank; Stratified by renal function (adequate vs borderline),tumor stage(T2N0vs >T2N0), PDL1 status(high vs low/negative); Hazard Ratio (HR) = 0.75, 98.457% CI 2-sided [0.563 to 0.985]; 95% CI: 0.594 to 0.934

6. Secondary Outcome: Metastasis-free Survival Per Investigator Assessment or Local Biopsy Review.
Description: MFS is defined as the time from date of randomization until the first recognition of distant metastases or death, whichever occurs first
Time Frame: Up to 48 months
Population: The full analysis set (FAS) Intention to treat included all randomized patients.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 533 | 530
Months | NA [24.2 to NA] — Median MFS was not reached due to insufficient number of participants with events 75th percentile MFS was not reached due to insufficient number of participants with events. | NA [15 to NA] — Median MFS was not reached due to insufficient number of participants with events 75th percentile MFS was not reached due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Durvalumab + Gemcitabine + Cisplatin vs Gemcitabine + Cisplatin; Test type: Superiority; p = 0.0002, Log Rank; Stratified by renal function(adequate vs borderline),tumor stage(T2N0 vs >T2N0), PDL1 status(high vs low/negative); Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.541 to 0.826] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Disease-specific Survival Per Investigator Assessment or Local Biopsy Review.
Description: DSS is defined as the time from the date of randomization until death due to bladder cancer
Time Frame: Up to 48 months
Population: The full analysis set (FAS) Intention to treat included all randomized patients.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 533 | 530
months | NA [NA to NA] — Median DSS was not reached due to insufficient number of participants with events 25th and 75th percentile DSS were not reached due to insufficient number of participants with events. | NA [50.9 to NA] — Median DSS was not reached due to insufficient number of participants with events 75th percentile DSS was not reached due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Durvalumab + Gemcitabine + Cisplatin vs Gemcitabine + Cisplatin; Test type: Superiority; p = 0.0081, Log Rank; Stratified by renal function(adequate vs borderline),tumor stage(T2N0 vs >T2N0), PDL1 status(high vs low/negative); Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.516 to 0.907] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Immunogenicity of Durvalumab When Used in Combination With Gemcitabine/Cisplatin as Measured by Presence of Antidrug Antibodies (ADA)
Description: Whole blood samples for assessing ADA for durvalumab in serum were collected from patients undergoing durvalumab treatment, following the specified assessment schedule. ADA prevalence is the proportion of patients with a positive ADA result at any time, baseline or post-baseline. Treatment-emergent ADA includes both treatment-induced and treatment-boosted ADA. Its incidence is the proportion of patients with treatment-emergent ADA positivity. Treatment-boosted ADA refers to a baseline-positive ADA titer that increased ≥4-fold during the study. Persistently positive patients have at least two post-baseline ADA-positive readings, with at least 16 weeks between the first and last, or an ADA-positive result at the final assessment. This includes baseline-positive patients meeting these criteria. Transiently positive is defined by at least one post-baseline ADA-positive reading without being persistently positive, including baseline-positive patients meeting these terms.
Time Frame: Up to 12 months
Population: The ADA analysis set includes all participants who had non-missing baseline ADA and at least one non-missing post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 453
Participants
  ADA positive at any visit (ADA prevalence) | 37
  Treatment-emergent ADA positive (ADA Incidence) | 8
  Treatment-boosted ADA | 1
  Treatment-induced ADA (Positive Post-baseline only) | 7
  ADA Positive at Baseline only | 29
  ADA Positive Post-baseline and Positive at Baseline | 1
  Persistently Positive | 4
  Transiently Positive | 4
  nAb Positive at any visit | 6

ADVERSE EVENTS:
Time Frame: Includes AEs between date of first dose and the earliest of: maximum date of (last dose or surgery) + 90days, date of first dose of subsequent anti-cancer therapy. Total follow up about 2 years. The frequency assessment was: Neoadjuvant, every 3 weeks, Post Surgery, every week, Adjuvant and Follow Up: every 4 weeks. All-cause mortality (death due to any cause): from randomization up to EFS IA2 DCO (April 29, 2024). Maximum timeframe of approximately 5.4 years.
Arm/Group | Durvalumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
All-Cause Mortality (participants affected / at risk) | 27/533 | 29/526
Serious Adverse Events (participants affected / at risk) | 326/530 | 287/526
Other Adverse Events (participants affected / at risk) | 522/530 | 511/526
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + Gemcitabine + Cisplatin (N=530) | Gemcitabine + Cisplatin (N=526)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (3) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (2)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1) | 1 (1)
Fungal endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Fungal peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Haematological infection (Infections and infestations) | 0 (0) | 1 (1)
Infected lymphocele (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 2 (2) | 2 (2)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Perinephric abscess (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 12 (12) | 5 (6)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 2 (2)
Postoperative wound infection (Infections and infestations) | 2 (2) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 19 (26) | 23 (28)
Pyelonephritis acute (Infections and infestations) | 6 (7) | 4 (4)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 1 (1)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 19 (20) | 14 (15)
Septic shock (Infections and infestations) | 8 (8) | 5 (5)
Severe acute respiratory syndrome (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Suspected covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 59 (80) | 69 (90)
Urosepsis (Infections and infestations) | 20 (22) | 10 (11)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (3) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative ileus (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rectal injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Stenosis of vesicourethral anastomosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Urethral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary tract injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 6 (6) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Candida test positive (Investigations) | 1 (1) | 0 (0)
Gastrointestinal stoma output increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 3 (3)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 6 (6) | 5 (5)
Sars-cov-2 test positive (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 17 (18)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hamartoma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 35 (35) | 27 (27)
Prostate cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Prostate cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 (21) | 10 (10)
Prostate cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 3 (3)
Cranial nerve palsies multiple (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic coma (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Iiird nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 2 (2)
Seizure (Nervous system disorders) | 1 (1) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 5 (5) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 25 (26) | 24 (29)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder wall calcification (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 4 (4)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 3 (4)
Hydronephrosis (Renal and urinary disorders) | 15 (17) | 8 (8)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 3 (3) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Obstructive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Perinephric collection (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 8 (8) | 10 (10)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (2)
Renal impairment (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal pelvis fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 3 (4)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3) | 2 (2)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract inflammation (Renal and urinary disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 4 (4) | 2 (2)
Vesicourethral fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Orchitis noninfective (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Prostatic dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8) | 9 (9)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 5 (5)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aortic occlusion (Vascular disorders) | 0 (0) | 1 (1)
Arterioenteric fistula (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 4 (4)
Distributive shock (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 5 (6) | 0 (0)
Femoral artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Lymphocele (Vascular disorders) | 7 (7) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (2)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fistula of small intestine (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 7 (7) | 4 (4)
Ileus paralytic (Gastrointestinal disorders) | 3 (4) | 2 (2)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 5 (5)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal strangulation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 6 (8) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 1 (1)
Asthenia (General disorders) | 0 (0) | 4 (6)
Death (General disorders) | 3 (3) | 5 (5)
Dehiscence (General disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 4 (4)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 3 (4) | 2 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 2 (2)
Bacterial abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bacteroides bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 9 (9) | 5 (5)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + Gemcitabine + Cisplatin (N=530) | Gemcitabine + Cisplatin (N=526)
Urinary tract infection (Infections and infestations) | 124 (181) | 108 (158)
Procedural pain (Injury, poisoning and procedural complications) | 46 (49) | 38 (43)
Alanine aminotransferase increased (Investigations) | 46 (65) | 38 (48)
Amylase increased (Investigations) | 34 (43) | 19 (26)
Blood creatinine increased (Investigations) | 94 (131) | 76 (97)
Lipase increased (Investigations) | 39 (49) | 27 (32)
Neutrophil count decreased (Investigations) | 80 (121) | 72 (102)
Platelet count decreased (Investigations) | 35 (48) | 32 (43)
Weight decreased (Investigations) | 41 (41) | 27 (28)
White blood cell count decreased (Investigations) | 28 (47) | 35 (58)
Decreased appetite (Metabolism and nutrition disorders) | 140 (196) | 131 (175)
Anaemia (Blood and lymphatic system disorders) | 200 (257) | 200 (239)
Hyperglycaemia (Metabolism and nutrition disorders) | 29 (33) | 23 (24)
Hyperkalaemia (Metabolism and nutrition disorders) | 44 (58) | 26 (30)
Hypokalaemia (Metabolism and nutrition disorders) | 31 (47) | 23 (34)
Hypomagnesaemia (Metabolism and nutrition disorders) | 56 (77) | 55 (73)
Arthralgia (Musculoskeletal and connective tissue disorders) | 54 (65) | 35 (39)
Back pain (Musculoskeletal and connective tissue disorders) | 50 (57) | 46 (54)
Myalgia (Musculoskeletal and connective tissue disorders) | 32 (35) | 13 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (27) | 28 (31)
Tinnitus (Ear and labyrinth disorders) | 36 (41) | 43 (48)
Dizziness (Nervous system disorders) | 42 (59) | 39 (43)
Hyperthyroidism (Endocrine disorders) | 30 (31) | 9 (10)
Dysgeusia (Nervous system disorders) | 40 (42) | 33 (38)
Headache (Nervous system disorders) | 59 (74) | 59 (69)
Neuropathy peripheral (Nervous system disorders) | 32 (40) | 29 (32)
Insomnia (Psychiatric disorders) | 43 (49) | 45 (56)
Hypothyroidism (Endocrine disorders) | 60 (64) | 11 (11)
Dysuria (Renal and urinary disorders) | 28 (33) | 19 (20)
Abdominal distension (Gastrointestinal disorders) | 28 (29) | 23 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (40) | 24 (30)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 (55) | 19 (20)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 41 (66) | 50 (66)
Alopecia (Skin and subcutaneous tissue disorders) | 49 (50) | 57 (58)
Pruritus (Skin and subcutaneous tissue disorders) | 80 (96) | 38 (42)
Rash (Skin and subcutaneous tissue disorders) | 67 (81) | 30 (34)
Hypertension (Vascular disorders) | 61 (71) | 42 (45)
Abdominal pain (Gastrointestinal disorders) | 65 (80) | 39 (45)
Abdominal pain upper (Gastrointestinal disorders) | 30 (38) | 22 (24)
Constipation (Gastrointestinal disorders) | 204 (276) | 201 (276)
Diarrhoea (Gastrointestinal disorders) | 106 (137) | 74 (88)
Dyspepsia (Gastrointestinal disorders) | 48 (55) | 47 (50)
Leukopenia (Blood and lymphatic system disorders) | 31 (52) | 37 (58)
Neutropenia (Blood and lymphatic system disorders) | 136 (212) | 163 (274)
Nausea (Gastrointestinal disorders) | 281 (425) | 254 (403)
Vomiting (Gastrointestinal disorders) | 101 (141) | 96 (138)
Asthenia (General disorders) | 93 (119) | 92 (120)
Thrombocytopenia (Blood and lymphatic system disorders) | 55 (75) | 55 (82)
Fatigue (General disorders) | 190 (269) | 169 (225)
Malaise (General disorders) | 34 (45) | 25 (32)
Oedema peripheral (General disorders) | 45 (55) | 45 (52)
Pyrexia (General disorders) | 107 (140) | 84 (113)
Hydronephrosis (Renal and urinary disorders) | 18 (19) | 29 (32)
Covid-19 (Infections and infestations) | 21 (23) | 30 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT03732677/Prot_002.pdf
  • Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT03732677/SAP_003.pdf